CLINICAL TRIAL: NCT00533416
Title: A Pilot Study of the Safety and Activity of Escalating Doses of ON 01910.Na in Patients With RAEB-1 AND RAEB-2 Myelodysplastic Syndrome (MDS) and AML With Trisomy 8
Brief Title: Safety of ON 01910.Na in Patients With Myelodysplasia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070225; 07-H-0225
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-04-27

CONDITIONS: Myelodysplastic Syndrome (MDS)
Keywords: Myelodyplastic Syndrome (MDS); Selective Mitotic Inhibitor; Targeted Therapy; Myelodysplastic Syndrome; MDS
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — ON 01910

INTERVENTIONS:
Drug: ON 01910 Na

SUMMARY:
This study will determine the highest dose of the experimental drug ON 01910.Na that can safely be given to patients with the bone marrow disorder myelodysplasia (MDS) and patients with refractory AML with trisomy 8. In this disease, the bone marrow can make some blood cells, but very few of these cells are released into the blood for use in the body. ON 01910.Na is an experimental drug that inhibits a protein called cyclinD1that is important for keeping MDS cells alive. In laboratory experiments, ON 01910.Na has acted against cyclinD1, causing MDS cells to die. The study will also evaluate how the body handles ON 01910.Na, the effect of the drug on MDS and AML and its side effects.

Patients 18 to 85 years old with MDS or AML who do not have a suitable sibling donor for a marrow transplant or who are not willing to have a transplant may be eligible for this study.

Participants receive ON 01910.Na in 2-week treatment cycles, with 3 to 5 days of drug infusion through a vein followed by 9 to 11 days of observation. To find the highest safe dose of ON 01910.Na, the first person enrolled in the study is given the smallest study dose of the drug for 3 days, followed 2 weeks later with a second dose for 3 days. If these doses are found safe, the next two people receive the same dose. If these subjects do well, the next group of patients receives the next higher dose level. The dose continues to be increased in groups of 3 to 6 subjects until the fourth and highest dose level is reached. Patients who do well on the treatment may receive an additional six cycles of ON 01910.Na (3 to 5 days of infusion once every other week for 12 weeks).

Before, during and after the treatment period, patients are periodically evaluated and monitored with the following tests and procedures:

* Physical examination and review of medical and medication history.
* Blood and urine tests.
* Pregnancy test for women of childbearing age.
* Electrocardiogram (EKG) and chest X-ray.
* Bone marrow biopsy.

DETAILED DESCRIPTION:
The myelodysplastic syndromes (MDS) and acute myelogenous leukemias (AML) are a group of heterogeneous diseases with wide variation in clinical presentation and disease severity. Typically patients are older adults with co-morbidities. AML and MDS are characterized by variable degrees of cytopenias (anemia, neutropenia, thrombocytopenia) due to ineffective hematopoiesis and dysplastic bone marrow morphology or hematological malignancy.

Treatment of MDS is unsatisfactory: chemotherapy has a limited role in the management of leukemic progression; autologous stem cell transplantation does not prolong relapse-free survival and stem cell transplantation is poorly tolerated in older individuals. Some MDS patients have been shown to respond to a wide variety of immunosuppressive agents ranging from corticosteroids to cyclosporine (CsA) and horse antithymocyte globulin (h-ATG). However, the overall response rate is less than 30% and relapse continues to be a problem. Few treatments appear to change the natural history of MDS however, growth factors, decitabine, and lenalidomide can improve cytopenias, and 5-azacytidine, can reduce transfusion requirements, and improve quality of life when compared to supportive care. In addition most MDS patients are older and tolerate aggressive therapies poorly.

Some AML patients can be cured with chemotherapy or by allogeneic stem cell transplantation. However standard treatment approaches are not effective for patients who become refractory to chemotherapy, elderly patients, and those who relapse after transplantation.

The management of MDS and relapsed/refractory AML patients therefore remains unsatisfactory and targeted therapies are needed. One such investigational drug, ON 01910.Na, is a potent inhibitor of cyclin D1 and mitosis. ON01910.Na shows activity against a broad spectrum of tumor cell lines. Animal model studies show little toxicity with a high therapeutic index in these tumors. In addition, the fact that MDS bone marrow (particularly trisomy 8) and patients with AML with the trisomy 8 abnormality (Sloand, unpublished data) over-express cyclin D1 and in vitro studies have demonstrated activity against cytogenetically abnormal cells and blasts despite minimal inhibition of normal hematopoiesis provides a rationale for its use in select patients with MDS or AML.

We therefore propose a non-randomized, pilot, dose escalating Phase I study of ON 01910.Na in MDS and patients with refractory AML with trisomy 8.

The primary objective is to determine the safety (including the maximum tolerated dose and/or dosing regimen) of ON 01910.Na when administered in escalating doses in select patients with MDS or AML. Secondary objectives include plasma pharmacokinetics and biological effects of ON 01910.Na on cell-cycle pathways of MDS or AML cells, and bone marrow RNA analysis to assess if gene expression can predict clinical response to ON 01910.Na in subjects with MDS.

The primary endpoint will be the toxicity profile at each dose level. Secondary endpoints will include the evaluation of early evidence of disease response by blast and cytogenetic improvement.

ELIGIBILITY:
* All patients 18-85 years old with RAEB1 or RAEB 2 MDS or refractory AML with trisomy 8 who lack a suitable matched sibling marrow will be considered for enrollment. Patients who have a suitable matched sibling donor will be referred for consideration of allogeneic bone marrow transplantation. Patients not willing to undergo transplantation or have relapsed following transplantation will be considered for protocol participation.

INCLUSION CRITERIA:

1. Histologically documented or cytologically confirmed diagnosis of MDS with WHO classification of RAEB-1 or 2 or Intermediate to High IPSS risk group.

   OR

   Refractory acute myelogenous leukemia (AML) with trisomy 8
2. Anemia requiring transfusion support with at least one unit of packed red blood cells per month for greater than or equal to 2 months

   OR

   Anemia (hemoglobin less than 9 or a reticulocyte count less than 60,000/microL)

   OR

   thrombocytopenia (platelet count less than 50,000/microL)

   OR

   neutropenia (absolute neutrophil count less than 500/microL).
3. Failed to respond to, relapsed following, or opted not to participate in bone marrow transplantation or other standard of care treatment options.
4. ECOG Performance Status of 0, 1, or 2.
5. Off all other treatments for MDS or AML (except filgrastim (G-CSF), erythropoietin, and transfusion support and related medications) for at least four weeks. Filgrastim (G-CSF) can be used before, during and after the protocol treatment for patients with documented neutropenia (less than 500/microL) as long as they meet the criteria for anemia and/or thrombocytopenia as stated above. Post transplant patients may continue to receive DLIs as needed.
6. Ages 18-85.

EXCLUSION CRITERIA:

1. Active infection not adequately responding to appropriate therapy.
2. Hypoplastic MDS (cellularity less than 10 percent) or an absolute neutrophil count of less than 200 cells/microL.
3. Active malignant disease (excluding non-melanoma skin carcinoma) other than AML.
4. Uncontrolled intercurrent illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
5. An expected survival, in the opinion of the investigator that would not permit a sufficient observation period for evaluating ON 01910.Na.
6. HIV positive patients.
7. Total bilirubin greater than 1.5 mg/dL not related to hemolysis or Gilbert s disease.
8. Serum creatinine greater than 1.5 mg/dL, or a calculated creatinine clearance of less than 60 mL/min/1.73 m(2).
9. Ascites requiring active medical management including paracentesis, peripheral bilateral edema, hyponatremia (serum sodium less than 134 meq/L.
10. Currently receiving any other investigational agents or concurrent chemotherapy, radiotherapy, or immunotherapy.
11. Current pregnancy, unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential or currently breastfeeding. Pregnant and nursing women are excluded from this study.
12. Psychiatric illness/social situations that would limit the patient s ability to tolerate and/or comply with study requirements.
13. Unable to understand the investigational nature of the study or give informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-09-14; Primary Completion 2012-06-04 (Actual); Study Completion 2012-06-04 (Actual)

PRIMARY OUTCOMES:
The toxicity profile at each dose level.

SECONDARY OUTCOMES:
Plasma pharmacokinetics, pharmacodynamics, and biological effects of hematologic improvement at each dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barrett J, Saunthararajah Y, Molldrem J. Myelodysplastic syndrome and aplastic anemia: distinct entities or diseases linked by a common pathophysiology? Semin Hematol. 2000 Jan;37(1):15-29. doi: 10.1016/s0037-1963(00)90027-1. PMID 10676908
- [Background] Toyama K, Ohyashiki K, Yoshida Y, Abe T, Asano S, Hirai H, Hirashima K, Hotta T, Kuramoto A, Kuriya S, et al. Clinical implications of chromosomal abnormalities in 401 patients with myelodysplastic syndromes: a multicentric study in Japan. Leukemia. 1993 Apr;7(4):499-508. PMID 8464227
- [Background] de Witte T, Suciu S, Verhoef G, Labar B, Archimbaud E, Aul C, Selleslag D, Ferrant A, Wijermans P, Mandelli F, Amadori S, Jehn U, Muus P, Boogaerts M, Zittoun R, Gratwohl A, Zwierzina H, Hagemeijer A, Willemze R. Intensive chemotherapy followed by allogeneic or autologous stem cell transplantation for patients with myelodysplastic syndromes (MDSs) and acute myeloid leukemia following MDS. Blood. 2001 Oct 15;98(8):2326-31. doi: 10.1182/blood.v98.8.2326. PMID 11588026
- [Derived] Olnes MJ, Shenoy A, Weinstein B, Pfannes L, Loeliger K, Tucker Z, Tian X, Kwak M, Wilhelm F, Yong AS, Maric I, Maniar M, Scheinberg P, Groopman J, Young NS, Sloand EM. Directed therapy for patients with myelodysplastic syndromes (MDS) by suppression of cyclin D1 with ON 01910.Na. Leuk Res. 2012 Aug;36(8):982-9. doi: 10.1016/j.leukres.2012.04.002. Epub 2012 Apr 21. PMID 22524974